CLINICAL TRIAL: NCT07255235
Title: Comparative Evaluation of C-Mac, Pentax Video Laryngoscopes, and Macintosh Laryngoscope in Endotracheal Intubation in Intensive Care Unit Wearing a Face Shield.
Brief Title: Comparison Between C-mac,Pentax Video Laryngoscopes and Machintosh Laryngoscope
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mai Mahmoud Mohamed Ali Mosa, Principle investigator, Minia University
Other Study IDs: 1463
Record Dates: First submitted 2025-04-24; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Intubation; Difficult or Failed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- C-mac video laryngoscope group: Endotracheal intubation will be performed using the C-Mac video laryngoscope under ICU conditions, while wearing a face shield. The procedure aims to assess time to intubation, ease of use, and success rate.
- Pentax video-laryngoscope group: Endotracheal intubation will be performed using the Pentax video laryngoscope under ICU conditions, while wearing a face shield. The procedure aims to assess time to intubation, ease of use, and success rate.
- Machintosh laryngoscope group: Endotracheal intubation will be performed using the traditional Macintosh laryngoscope under ICU conditions, while wearing a face shield. The procedure aims to assess time to intubation, ease of use, and success rate.

SUMMARY:
Asses and compare the practility and the level of difficulty in using C-mac and pentax video-laryngoscopes or the traditional Macintoch laryngoscope in intubation in ICU patients while wearing face shield

DETAILED DESCRIPTION:
The endotracheal intubation will be performed with anesthesiologist working in ICU previously trained and experienced in videolaryngoscopy and will be classified according to their skill into 3 groups: Junior (1 year up to 3 year) senior, (3 year up to 8 years) and consultant (more than 8 years) experience. All the laryngoscopist groups will equally attend in performing intubation of the studied group. After the patient consent, the allocation will be opened and preparation for intubation will start. All the intubations will be performed with the presence of two laryngoscopist: one of them at least senior or consultant. After confirmation of well working standard monitoring (ECG, blood pressure, Spo2 and End-tidal CO2) and preoxygenation with 100% oxygen, induction with propofol (1-2 mg/kg) and rocuronium (0.9 mg/kg) will be achieved by an assistant.

While wearing head-fitted face shield, the anesthetist will perform intubation with suitable sized laryngoscopy blade and endotracheal tube. Successful placement of ETT will be confirmed by both auscaltation and capnography (normal appearing waveform over four or more breathing cycles). During endotracheal intubation, anesthesiologists will be permitted to make ergonomic adjustments, such as altering the bed height, position of the patient head and utilize external laryngeal manipulations, equipment adjustment and use of stylet based on their personal preferences. After three failed attempts of intubation, alternative techniques will be used and subsequently, they will not be included in the analysis. Alternative techniques such as gum elastic bougie, laryngeal mask airway (LMA), Cricothyrotomy set will be ready to any unexpected difficult airway. An intubation attempt is defined as introduction of laryngoscope and its subsequent removal with or without endotracheal tube (ETT) placement. Correct placement of ETT in first attempt by an individual laryngoscopist will be defined as first-pass successful intubation.

ELIGIBILITY:
Inclusion Criteria:

* All patients between age 18 - 65 year who will need elective orotracheal intubation will be included in the study after collection of data relevant to intubation

Exclusion Criteria:

* • Patients with BMI > 35.

  * Pregnant and lactating patients.
  * Burn and facial trauma patients.
  * Suspected or confirmed spine injury.
  * Presence of any predictors or history of difficult intubation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients between age 18 - 65 year who will need elective orotracheal intubation will be included in the study after collection of data relevant to intubation except:
  * Patients with BMI > 35.
  * Pregnant and lactating patients.
  * Burn and facial trauma patients.
  * Suspected or confirmed spine injury.
  * Presence of any predictors or history of difficult intubation.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Success rate of first pass of orotracheal intubation | Untill the end of the study in average of 1 year
  Passage of the orotracheal tube from the first time confirmed By capnography

CONTACTS AND LOCATIONS:
Overall Officials: Mai M Mohamed Ali, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine Minia University, Ma‘şarat Samālūţ, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taboada M, Almeida X, Carinena A, Costa J, Carmona-Monge J, Agilda A, Barreiro L, Castillo J, Williams K, Segurola J, Alvarez J, Seoane-Pillado T. Complications and degree of difficulty of orotracheal intubation in the Intensive Care Unit before and after the establishment of an intubation protocol for critically ill patients: a prospective, observational study. Rev Esp Anestesiol Reanim (Engl Ed). 2024 Jan;71(1):17-27. doi: 10.1016/j.redare.2023.12.004. Epub 2023 Dec 15. PMID 38104962
- [Result] Vig S, Bhan S, Gupta N, Meena JK, Bhatnagar S. Comparison of Mc Grath-MAC and C-MAC video laryngoscopes for intubation in a COVID simulated mannequin by novice users wearing face protective gear: A randomized crossover trial. Saudi J Anaesth. 2021 Apr-Jun;15(2):131-136. doi: 10.4103/sja.sja_1058_20. Epub 2021 Apr 1. PMID 34188630